CLINICAL TRIAL: NCT02998320
Title: Evaluation of Compliance With Treatment by Elvitegravir/Cobicistat/FTC/Tenofovir Alafenamide (E/C/F/TAF) in HIV Post-exposure Prophylaxis (to Infected Blood or Sexual Contact)
Brief Title: Evaluation of Compliance With Treatment by Genvoya in HIV Post-exposure Prophylaxis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe d'Etude sur le Risque d'Exposition des Soignants aux Agents Infectieux (Network)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEFR1044015
Record Dates: First submitted 2016-12-14; First posted 2016-12-20 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: HIV Risk
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genvoya (Experimental): Genvoya (E/C/F/TAF) Tablet (oral use) : 150/150/200/10 mg, one tablet each day for 28 days
  Interventions: Drug: Genvoya

INTERVENTIONS:
Drug: Genvoya — Oral use (one tablet each day); 150/150/200/10 mg; 28 days
  Other Names: (E/C/F/TAF) ATC Code: J05AR18

SUMMARY:
This study measures the proportion of enrolled patients taking the uninterrupted HIV post-exposure prophylaxis Genvoya for four weeks

DETAILED DESCRIPTION:
This study measures the proportion of enrolled patients taking the uninterrupted HIV post-exposure prophylaxis Elvitegravir/Cobicistat/FTC/Tenofovir alafenamide (E/C/F/TAF) for four Weeks.

Elvitegravir is an HIV-1 integrase strand transfer inhibitor (INSTI). Cobicistat is a selective, mechanism-based inhibitor of cytochrome P450 (CYP) enzymes of the CYP3A subfamily. Emtricitabine is a nucleoside reverse transcriptase inhibitor (NRTI) and nucleoside analogue àf 2'-dexicytidine. Tenofovir alafenamide is a nucleotide reverse transcriptase inhibitor (NtRTI) and phosphonoamidate prodrug of tenofovir (2'-deoxyadenosine monophosphate analogue).

ELIGIBILITY:
Inclusion Criteria:

* an age above 18 years
* consultation within 48 hours following a risk of HIV transmission (blood or sexual contact)
* indication for HIV post-exposure prophylaxis (according to French guidelines)
* person able to understand the nature of the study
* person who signed his consent form to participate in the study

Exclusion Criteria:

* person exposed to HIV risk from person infected by HIV, whose therapeutic history justifies the prescription of another combination of antiretroviral drugs
* contraindications to the prescription of Genvoy
* other medical contraindications
* person infected by hepatitis B virus
* pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients taking the uninterrupted HIV post-exposure prophylaxis for four weeks | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: David Rey, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (16):
- France (16):
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Saint-André, Bordeaux
  - CHU Ambroise Paré, Boulogne-Billancourt
  - Hôpital Manchester, Charleville-Mézières
  - CHU Dijon, Dijon
  - Hôpital Croix Rousse, Lyon
  - CHR de Metz, Metz
  - CHU Bichat, Paris
  - Hôpital Tenon, Paris
  - Hôpital Saint-Antoine, Paris
  - GH Pitié Salpetriere, Paris
  - CHU de Reims, Reims
  - CHU, Rennes
  - Hôpitaux Universitaires, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpital de Tourcoing, Tourcoing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gantner P, Hessamfar M, Souala MF, Valin N, Simon A, Ajana F, Bouvet E, Rouveix E, Cotte L, Bani-Sadr F, Hustache-Mathieu L, Lebrette MG, Truchetet F, Galempoix JM, Piroth L, Pellissier G, Muret P, Rey D; E/C/F/TAF PEP Study Group. Elvitegravir-Cobicistat-Emtricitabine-Tenofovir Alafenamide Single-tablet Regimen for Human Immunodeficiency Virus Postexposure Prophylaxis. Clin Infect Dis. 2020 Feb 14;70(5):943-946. doi: 10.1093/cid/ciz577. PMID 31804669